CLINICAL TRIAL: NCT07082673
Title: Efficacy and Tolerability of a Food Supplement Based on a Sea Buckthorn (Hippophae Rhamnoides L.) Extract Taken at Two Different Doses for the Management of Balance in Bowel Function in Subjects With Primary Functional Constipation: Single-center, Randomized, Placebo-controlled, Parallel-arm, Double-blind Clinical Trial
Brief Title: The Beneficial Effect on the Bowel Function of a Food Supplement Based on Sea Buckthorn (Hippophae Rhamnoides L.) Extract in Subjects With Primary Functional Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ISTITUTO FARMOCHIMICO FITOTERAPICO: EPO SRL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OLIVGUT2501
Record Dates: First submitted 2025-07-15; First posted 2025-07-24 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Functional Constipation (FC)
Keywords: Functional constipation; Food supplement; sea buckthorn; Hippophae rhamnoides L.

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, placebo-controlled, parallel-arm, double-blind clinical trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP 1: subjects who will take the dietary supplement based on sea buckthorn extract 500 mg dose. (Experimental): GROUP 1: subjects who will take the dietary supplement based on sea buckthorn extract (Hippophae rhamnoides L.) at a dose of 500 mg - DOSE A (1 capsule of supplement + 2 capsules of placebo).
  Interventions: Dietary Supplement: Sea Buckthorn (Hippophae rhamnoides L.) botanical extract 500 mg.
- GROUP 2 subjects who will take the food supplement based on sea buckthorn 1500 mg dose. (Experimental): GROUP 2 subjects who will take the food supplement based on sea buckthorn (Hippophae rhamnoides L.), at a dose of 1500 mg - DOSE B (3 capsules of supplement).
  Interventions: Dietary Supplement: Sea buckthorn (Hippophae rhamnoides L.) 1500 mg.
- GROUP 3 subjects who will take placebo. (Placebo Comparator): GROUP 3 subjects who will take placebo (3 capsules of placebo).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sea Buckthorn (Hippophae rhamnoides L.) botanical extract 500 mg. — Dietary supplement based on sea buckthorn extract (Hippophae rhamnoides L.) at a dose of 500 mg - DOSE A (1 capsule of supplement + 2 capsules of placebo).
  Arms: GROUP 1: subjects who will take the dietary supplement based on sea buckthorn extract 500 mg dose.
Dietary Supplement: Sea buckthorn (Hippophae rhamnoides L.) 1500 mg. — Dietary supplement based on sea buckthorn (Hippophae rhamnoides L.), at a dose of 1500 mg - DOSE B (3 capsules of supplement).
  Arms: GROUP 2 subjects who will take the food supplement based on sea buckthorn 1500 mg dose.
Dietary Supplement: Placebo — Placebo (3 capsules of placebo).
  Arms: GROUP 3 subjects who will take placebo.

SUMMARY:
The study will aim to evaluate the efficacy and tolerability of a supplementation with Sea Buckthorn (Hippophae rhamnoides L.) at two different dosages for the management of the balance of intestinal function in subjects with primary functional constipation.

The primary outcome is the improvement of the frequency of bowel movements (SCBM) in subjects with functional constipation; then the secondary outcomes are the 1) improvement in stool consistency, assessed through the Bristol Stool Form Scale (BSFS) and 2) reduction in the typical symptoms of constipation, such as feeling of bloating and abdominal distension, feeling of heaviness, abdominal pain and flatulence, improving the quality of life of the subjects affected by primary functional constipation.

DETAILED DESCRIPTION:
This study aims to understand if a food supplement based on sea buckthorn extract (Hippophae rhamnoides L.) can be useful for managing primary functional constipation.

Sea buckthorn is a plant known for having positive effects on bowel regularity. In fact, it is present in the plant list of the Italian Ministry of Health that allows its use in food supplements for this property. Sea buckthorn has long been used in various parts of the world for its beneficial properties and contains many nutrients and active substances. In particular, several studies have suggested that sea buckthorn could improve intestinal motility. In addition, it seems that it can increase the production of a protein that helps transport water in the intestine, softening the stool, similar to osmotic laxatives.

The study involves the recruitment of a total of 135 participants, who will be divided into three parallel groups, with 45 subjects per group. It is a "blind" and placebo-controlled study, which means that the participants will be divided randomly, and no one (neither the participants nor the doctors) will know who will take the real supplement and who will take an inactive substance (placebo). The participants who will be included in the study are subjects of both sexes, aged between 18 and 70 years, who must have symptoms of chronic constipation for at least 3 months, with an onset at least 6 months before enrollment in the study.

To be eligible to participate, the subjects must also meet specific criteria regarding stool frequency and stool consistency. Specifically, they must have fewer than three complete spontaneous bowel movements (SCBM) per week and present at least one of the following conditions in more than 25% of defecatory acts: lumpy or hard stools (BSFS type 1 or 2), sensation of incomplete evacuation, sensation of anorectal obstruction/blockage, or need for manual maneuvers to facilitate evacuation.

In addition, participants must not have predominant abdominal pain that occurs more than one day per week, thus excluding subjects with IBS-C.

Finally, participants must not take any type of medication for bowel function during the study, must test negative for HIV and, for women of childbearing age, for pregnancy. They must also be able to understand and sign the informed consent and comply with the protocol requirements.

The three groups of participants will receive the following treatments for the duration of the study:

* Group 1 (DOSE A): 45 subjects who will take the sea buckthorn food supplement at a dose of 500 mg (1 capsule of supplement + 2 capsules of placebo).
* Group 2 (DOSE B): 45 subjects who will take the sea buckthorn food supplement at a dose of 1500 mg (3 capsules of supplement).
* Group 3 (Placebo): 45 subjects who will take a placebo (3 capsules of placebo). Sea buckthorn extract has a significant history of consumption in the European Union and is considered a safe product, for which no adverse events related to the intake of the supplement are expected, including harm to the fetus in the case of pregnancy. However, participants will be continuously monitored, and in case of suspected adverse reactions, these will be reported via the online phytovigilance system VigiErbe (www.vigierbe.it). Although no adverse events are expected, the possibility of unexpected individual reactions to the active ingredients or excipients of the supplement or placebo cannot be completely ruled out, for this reason, in the event of unexpected serious adverse reactions (SUSAR), these will be reported to the Ethics Committee and noted in the CRF form.

As a precautionary measure, sexually active women of childbearing age will be required to use a contraceptive method during sexual intercourse for the entire duration of the study. If pregnancy occurs during the study, the participant will be excluded. On the other hand, if the supplement results to be effective, participants who take it (at one of the two doses) may experience an improvement in their bowel function, as well as benefit from relief from the main symptoms of constipation such as abdominal pain and bloating. This may also lead to a better quality of life.

The OLIVGUT25 study will be conducted at a single center: COMEGEN Soc. Coop. Sociale, located in Viale Maria Bakunin, 41 (Parco S. Paolo), 80126 - Naples. The Principal Investigator of the study is Dr. Matteo Laringe, also affiliated with COMEGEN Soc. Coop. Social.

Subjects enrolled in the study will be followed at this location for the duration of their participation.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 70 years
* able to understand and sign informed consent
* HIV negative test
* negative pregnancy test
* with symptoms of chronic constipation for at least 3 months (with onset at least 6 months earlier)
* absent/non-predominant abdominal pain that occurs less than one day per week and, therefore, not affected by IBS-C
* who have less than three SCBWs per week and at least one of the following conditions:

  * in more than 25%* of defecatory acts
  * lumpy or hard stools (BSFS type 1 or 2) in more than 25% of bowel movements
  * feeling of incomplete evacuation in more than 25% of defecations
  * feeling of anorectal obstruction/blockage in more than 25% of defecations
  * carry out manual manoeuvres to facilitate evacuation in more than 25% of defecations
* able to understand and comply with the requirements of the protocol

Exclusion Criteria:

* pregnancy
* lactation
* HIV positive
* do not meet inclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of the sea buckthorn-based dietary supplement in improving the frequency of Spontaneous Complete Bowel Movement (SCBM). | [Time frame: T0 (baseline), T1 (28 days of treatment)].
  Frequency of Spontaneous Complete Bowel Movement (SCBM), defined by EMA as an appropriate primary endpoint in the clinical evaluation of the efficacy of active ingredients for chronic functional constipation as it incorporates the concept of spontaneity without taking any salvage treatment (drugs or any other laxative, including dietary supplements, enemas or suppositories) within 24 hours before the bowel movement, as well as the completeness of the bowel movement.
  EVALUATION METHOD:
  Average value of the number of SCBMs/week in the previous month:
  1. referred by the subject at the recruitment visit (T0) and reported by the investigator physician on the patient record (Case Reporting Form - CRF), and
  2. calculated at the final visit (T1) on the basis of what the subject reported in the bowel function diary.

SECONDARY OUTCOMES:
Stool consistency, which together with the frequency of SCBM, has been indicated in the EMA and EFSA guidelines as an equally valid indicator of the condition of functional constipation. | [Time frame: T0 (baseline), T1 (28 days of treatment)].
  EVALUATION METHOD: Bristol Stool Form Scale (BSFS), a validated instrument that assesses stool consistency on a spectrum of seven types. Type 1 and 2 stools denote hard or lumpy stools, while type 6 and 7 stools are indicative of loose or watery stools. The stools that characterize subjects with constipation are type 1 or 2. The consistency of the stool, expressed by the Bristol Scale, will be: 1) reported by the subject at the recruitment visit (T0) and reported by the investigator physician on the patient record (Case Reporting Form - CRF), and 2) calculated at the final visit (T1) on the basis of what the subject reported in the bowel function diary.
Assessment of the characteristic symptoms of the constipated subject: Feeling of bloating and abdominal distension, Feeling of heaviness, Abdominal pain, Flatulence (Bowel Function Diary). | [Time frame: up to 28 days].
  Bowel Function diary (BF diary). The diary consists of:
  1. parts that the subject will need to fill out at the time of bowel evacuation (date and time, BSFS)
  2. parts that the subject will have to fill in every day, regardless of the occurrence of an SCBM, such as: the evaluation of the characteristic symptoms of the constipated subject (feeling of bloating and abdominal distension, feeling of heaviness, abdominal pain, flatulence), through the compilation of a 5-point Likert scale (1 no discomfort - 5 maximum discomfort),
  3. the possible use of "salvage treatment",
  4. recording of daily fluid intake.
  The extent of the symptoms, expressed through the 5-point Likert Scale, will be:
  1. reported by the subject at the recruitment visit (T0) and reported by the investigator physician on the patient record (Case Reporting Form - CRF), and
  2. calculated at the final visit (T1) on the basis of what the subject reported on the function diary.
Possible use of "salvage treatment". | [Time frame: up to 28 days].
  Entry in the bowel function diary (BF diary). Subjects will have to record in the diary the possible use of "salvage treatment" (drugs or any other laxative, including food supplements, enemas or suppositories) in order to improve intestinal function. Taking such treatments will not directly result in the exclusion of the subject from the study or the discontinuation of the investigational treatments, but whether or not the subject's data will be retained in the analysis of the results will be evaluated by the principal investigator. Subjects will be instructed prior to initiation of treatment on whether to take salvage treatment by the investigators. In particular, the intake of rescue treatments will be allowed if recorded in the diary and if the subject should incur a decrease of at least one SCBM per week.
Evaluation of the impact of constipation on perceived quality of life in the last 4 weeks. | [Time frame: T0 (baseline), T1 (28 days of treatment)].
  Quality of Life Questionnaire (Short Form Health Survey-12 -SF-12) was developed in a multi-year study of patients with chronic conditions. It is a validated questionnaire widely used in clinical practice for self-assessment of quality of life against a generic disorder.
  Quality of life will be assessed through the SF-12 questionnaire score:
  1. as reported by the subject at the recruitment visit (T0) and
  2. as reported by the subject at the final visit (T1).

CONTACTS AND LOCATIONS:
Locations (1):
- COMEGEN Soc. Coop. Sociale, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No